CLINICAL TRIAL: NCT01540214
Title: Prevalence of Overactive Bladder (OAB) in Patients With Pelvic Organ Prolapse (POP) and Predictors of Symptoms of OAB After Surgical Correction of POP
Brief Title: Study of Overactive Bladder in Women With Prolapse
Acronym: SOAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Astellas Pharma Inc (Industry); Continentie Stichting Nederland (Continence Foundation The Netherlands) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2011/456
Record Dates: First submitted 2012-02-10; First posted 2012-02-28 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2012-12

CONDITIONS: Urinary Bladder, Overactive; Pelvic Organ Prolapse
Keywords: Urinary Bladder, Overactive; Pelvic Organ Prolapse; Gynecologic Surgical Procedures; Urodynamics
MeSH Terms: conditions — Urinary Bladder, Overactive; Pelvic Organ Prolapse | interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- POP surgery: All women who present with POP at the outpatient clinic of our centre and who will undergo prolapse repair surgery will be asked informed consent for participation in this study
  Interventions: Other: Pre- and postoperative evaluations

INTERVENTIONS:
Other: Pre- and postoperative evaluations — At baseline before surgery and at 6 and 12 months after surgery: questionnaires, bladder diary, pelvic examination with additional ultrasound (one extra outpatient clinic visit at 6 months compared to standard care).
  At baseline before surgery and at 12 months after surgery: urodynamics with additional urine sampling (one extra outpatient clinic visit at 12 months compared to standard care).
  At time of surgery: additional cystoscopy.

SUMMARY:
Pelvic organ prolapse (POP) is a common problem. Symptoms of overactive bladder (OAB) are present in approximately 50% of patients with POP. For many women the accompanying symptoms of OAB are an important reason for seeking help for their POP. Surgical repair of prolapse may improve OAB complaints. Persisting or de novo OAB symptoms are strongly correlated with dissatisfaction with the final results of an operation for POP.

The primary aim of this research project is to investigate the difference in prevalence (i.e. improvement) of OAB and bothersome OAB symptoms at 6 and 12 months after POP repair surgery. The secondary objectives are to determine changes in bladder function at 6 and 12 months after surgery and to identify predictive factors for persistence, disappearance or de novo symptoms of OAB after POP surgery.

Women who present with POP and who will undergo surgical treatment will be evaluated at baseline before their surgery and will be followed for the duration of one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age 18 or greater, with a pelvic organ prolapse stage II to IV as defined by the POP-Q system
* Patient is a candidate for prolapse repair surgery (as based on history and physical examination)
* Patient is capable to fill out bladder diaries and questionnaires and understands the Dutch written and spoken language

Exclusion Criteria:

* Patients who currently use anticholinergic medication
* Patients with neurological causes of OAB
* Patients who are pregnant
* Patients with a history of cancer in the pelvic region, treated with radiotherapy or surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women who present with POP at the outpatient clinic of our centre and who will undergo prolapse repair surgery will be asked informed consent for participation in this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in prevalence of OAB as measured by bladder diary and validated disease specific questionnaires at 6 months | At baseline before surgery and at 6 months after surgery
The change from baseline of bothersome OAB symptoms as measured by bladder diary and validated disease specific questionnaires at 6 months | At baseline before surgery and at 6 months after surgery
  The bother of OAB symptoms, measured by validated disease specific questionnaires, will be presented by scores that reflect the degree of severity of the voiding dysfunction. The presence of bothersome OAB symptoms will be dichotomized in patients with symptoms and moderate to severe bother (symptomatic) and patients with absence of symptoms or with only little or no bother (asymptomatic).
The change from baseline in prevalence of OAB as measured by bladder diary and validated disease specific questionnaires at 12 months | At baseline before surgery and at 12 months after surgery
The change from baseline of bothersome OAB symptoms as measured by bladder diary and validated disease specific questionnaires at 12 months | At baseline before surgery and at 12 months after surgery
  The bother of OAB symptoms, measured by validated disease specific questionnaires, will be presented by scores that reflect the degree of severity of the voiding dysfunction. The presence of bothersome OAB symptoms will be dichotomized in patients with symptoms and moderate to severe bother (symptomatic) and patients with absence of symptoms or with only little or no bother (asymptomatic).

SECONDARY OUTCOMES:
Change from baseline in outcomes of urodynamic studies (presence of detrusor overactivity (DO), bladder outflow obstruction (BOO)) at 12 months | At baseline before surgery and at 12 months after surgery
Change from baseline in POP-Q stage at 6 and 12 months | At baseline before surgery, at 6 and 12 months after surgery
Change from baseline in outcomes of ultrasound assessment (bladder wall thickness, bladder neck descent, retrovesical angle) at 6 and 12 months | At baseline before surgery, at 6 and 12 months after surgery
Cystoscopic assessment of trabeculation | At time of surgery
Change from baseline in concentration of urinary biomarkers at 12 months | At baseline before surgery and at 12 months after surgery
  Concentration of urinary biomarkers: nerve growth factor (NGF), prostaglandin E2 (PGE2) and adenosine triphosphate (ATP) levels in urine normalized against creatinine concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Vierhout, MD, PhD, Principal Investigator — Radboud University Medical Center; John PF Heesakkers, MD, PhD, Principal Investigator — Radboud University Medical Center; Myrthe M Tijdink, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands